CLINICAL TRIAL: NCT00226252
Title: Manual Wheelchair Propulsion Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Pittsburgh Healthcare System (U.S. Federal Agency)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Michael Boninger, Chair, Department of Physical Medicine and Rehabilitation, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 02159
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Manual Wheelchair Users
Keywords: Wheelchair; Propulsion; Biomechanics
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Instruction Only (IO) (Experimental): IO participants will train on the dynamometer for the same length of time as the Feedback Group. They will only be instructed to follow what they learned from the video presented at the beginning of the training session.
  Interventions: Procedure: Instruction Only
- Instruction and Feedback Group (FB) (Experimental): The FB group will receive video training, and real time feedback from the SMART Wheel as they push their wheelchair. A monitor displaying a random combination and amount of biomechanical feedback variables will be placed in front of subjects. Subjects will be instructed to adjust their stroke to optimize their biomechanics with feedback from the screen.
  Interventions: Procedure: Instruction and Feedback
- Control Group (No Intervention): Wheelchair characteristics will be noted; however, no wheelchair manipulation or changes in equipment will be performed or recommended.

INTERVENTIONS:
Procedure: Instruction Only — Video details an individual propelling a manual wheelchair with biomechanically correct propulsion technique.
  Arms: Instruction Only (IO)
Procedure: Instruction and Feedback — Individuals will watch video of correct propulsion technique and will receive real-time feedback from the SMART Wheel as they push their wheelchair to help optimize their propulsion technique.
  Arms: Instruction and Feedback Group (FB)

SUMMARY:
The purpose of this research study is to investigate a manual wheelchair training program to improve the way manual wheelchair users push their wheelchairs.

DETAILED DESCRIPTION:
The purpose of this research is to create a manual wheelchair propulsion-training program (MWPTP) that emphasizes propulsion techniques that improve the manual wheelchair users stroke pattern and efficiency. It is our hope that the design of a manual wheelchair-training program can help to minimize the upper extremity pain and injury often associated with manual wheelchair propulsion.

The MWPTP will exist in three forms, and will be given to three randomly assigned groups of subjects. An instruction only group (IO) will receive general instructions on how to best propel their wheelchair. A feedback group (FB) will receive additional instruction in wheelchair propulsion using a monitor displaying a random combination and amount of biomechanical feedback variables, such as cadence and proportion of time spent in propulsion. Subjects will be coached to develop an appropriate propulsion style that minimizes all of the predetermined feedback measures, which indicate poor technique and maximize all of the graphical measures indicating good propulsion technique. A control group (CG) will receive only testing which will be identical to the testing procedures followed by the IO and FB groups.

Participation in this study will consist of four visits to the Human Engineering Research Lab (HERL) for the FB, IO and CG. Visits 1-4 will be the same, except visit 4 will not include training for any of the groups. All subjects will use their own wheelchair and cushion; however researchers will attach SMART Wheels TM to the subjects' wheelchair in place of their current wheels. The SMART Wheels TM are used to record the forces and moments that occur during propulsion and will not alter the dimensions or feel of the subjects current wheelchair. During each visit, all subjects will be asked to push over a real life course that includes various grades and surfaces. Then they will be asked to push on a wheelchair dynamometer at 1 meter/sec for one minute, 2 meter/sec for one minute, and a self selected speed for one minute. During this time, data will may also be collected with use of an Optotrak kinematic measurement system that incorporates a camera 3D-motion analysis system.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or greater
* Use of a manual wheelchair as primary means of mobility (>80% of their ambulation)
* Spinal Cord Injury (SCI) cervical 7 level and lower

Exclusion Criteria:

* Wheelchair athletes having competed in racing in the last year.
* Current upper limb pain that limits mobility.
* <1 year post inpatient rehabilitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2003-12; Primary Completion 2008-03 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Stroke frequency, peak forces, time spent in propulsion | initial visit, visit 2 (1 week later), visit 3 (2 weeks later), visit 4 (3 months from initial visit)
Stroke pattern | initial visit, visit 2 (1 week later), visit 3 (2 weeks later), and visit 4 (3 months from initial visit).

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Boninger, MD, Principal Investigator — University of Pittsburgh and VA Pittsburgh Healthcare System
Locations (1):
- Human Engineering Research Laboratories, Pittsburgh, Pennsylvania, United States